CLINICAL TRIAL: NCT04949243
Title: Rapid Acceleration for Diagnostics in Underserved Populations: Home Testing
Acronym: SYCT
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108149
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who use the self administered SARs-CoV-2 antigen testing kits
  Interventions: Behavioral: Behavioral questionaires

INTERVENTIONS:
Behavioral: Behavioral questionaires — Behavioral surveys and questionaires

SUMMARY:
This observational, cohort sub-studyis embedded within a larger public health intervention that distributes at-home, self-administered, SARS-CoV-2 antigen testing kits to households within pre-selected communitiesthrough the CDC.Within this sub-study, we will evaluate the socio-behavioral mechanisms of SARS-CoV-2 community transmission, including social interactions, health behaviors, healthcare utilization, knowledge, disease burden, and feasibility of at-home testing. The study hypothesis is that positive at-home test results will be associated withaltered self-reported social interactions and altered health behaviors compared to negative test results. Surveys and questionnaires will be completed by participants through the smartphone app or via call center phone calls according to the schedule of events.Questionnaires will collect data on demographic characteristics, medical history and health status, COVID testing and symptoms, social interactions, knowledge of prevention strategies, infection risk, and attitudes towards vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported primary residence within the pre-identified communities
2. Age> 8 years at enrollment
3. Provision of signed and dated informed consent form

Exclusion Criteria: None if above are met

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children > 8 years of age living within pre-identified communities participating in the public health intervention
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: christoph Hornik, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Greenville Pitt County, Greenville, North Carolina
  - Hamilton County, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The project team utilized a robust communications campaign and mobilized community partners to assist with outreach and to organize COVID-19 (SARs-CoV-2) antigen testing kit distribution events. Community members received tests via online order (distributed by Amazon), and in person at local distribution centers and events.
Groups:
- People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits: The observational sub-study was open to the general population of targeted counties, and embedded within the larger public health intervention that distributed at-home, self-administered COVID tests. The sub-study looked at potential socio-behavioral mechanisms of SARS-CoV-2 Community Transmission: social interactions, health behaviors, healthcare utilization, knowledge, disease burden, feasibility of at-home testing.
Period: Overall Study
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
Started | 338
Completed | 263
Not Completed | 75

BASELINE CHARACTERISTICS:
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
Number analyzed (Participants) | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.10 (14.37)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 226
  Sex: Male | 88
  Sex: Not Indicated | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 295
  Unknown or Not Reported | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 34
  White | 252
  More than one race | 13
  Unknown or Not Reported | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 338

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Not Following Social Distancing Guidelines
Description: Number of participants who reported at their first follow-up assessment as having close contact (within 6 feet) with people who do not live with them.
Time Frame: 2 weeks
Population: Data not collected on 116 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
Number analyzed (Participants) | 222
Participants | 164

2. Secondary Outcome: Number of Participants That Avoided Public Spaces, Gatherings, or Crowds as a Prevention Measure
Description: Number of participants who reported at their first follow-up assessment as having avoided public spaces, gatherings, or crowds as a prevention measure.
Time Frame: 2 weeks
Population: Data not collected on 114 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
Number analyzed (Participants) | 224
Participants | 84

3. Secondary Outcome: Number of Participants Who Are Knowledgeable of Precautionary Measures to Prevent Infection
Time Frame: 4 months
Population: Data not collected.
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Positive SARs-CoV-2 Antigen Test Results
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
Number analyzed (Participants) | 338
Participants | 7

5. Secondary Outcome: Number of Healthcare Utilization Measures
Time Frame: 4 months
Population: Data not collected.
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | People Who Use the Self Administered SARs-CoV-2 Antigen Testing Kits
All-Cause Mortality (participants affected / at risk) | 0/338
Serious Adverse Events (participants affected / at risk) | 0/338
Other Adverse Events (participants affected / at risk) | 0/338

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT04949243/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT04949243/ICF_000.pdf